CLINICAL TRIAL: NCT02003989
Title: Revealing Increased Axonal Loss in Treated HIV Patients
Acronym: OCTIHIV
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RBM_CLL_2012-7
Record Dates: First submitted 2013-11-29; First posted 2013-12-06 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-05

CONDITIONS: HIV Seropositivity
MeSH Terms: conditions — HIV Seropositivity | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients: HIV patients infected for more than ten years with undetectable viral load, undergoing ophthalmologic examination and MRI
  Interventions: Other: ophthalmologic examination and MRI
- control: non HIV patients (same gender and age) undergoing ophthalmologic examination and MRI
  Interventions: Other: ophthalmologic examination and MRI

INTERVENTIONS:
Other: ophthalmologic examination and MRI — thorough investigation of patients, not included in usual care.

SUMMARY:
HIV patients may suffer sooner from aging than average population, including brain aging. Our hypothesis is that if brain dysfunctions are explained by a quicker loss of neurons in HIV patients, this loss could be detected earlier by a thinning down of retinal nerve fiber layer (RNFL), compared to non HIV patients of the same age.

DETAILED DESCRIPTION:
The investigators aim to compare the thickness of the RNFL and the thickness of the RCGs measured by spectral domain OCT between patients infected by HIV and patients of same age non infected by HIV.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection known since at least 10 years
* viral load undetectable under ARV treatment since at least 5 years, whatever the type of ARV
* lymphocytes CD4 > 350, whatever the CD4 nadir
* signed informed consent

Exclusion Criteria:

* History of ocular pathology, eye surgery, or intraocular injection
* Familial History of glaucoma
* ametropia (>3 dioptres on the sphere and >1,5 dioptres on the cylinder)
* known neurological pathology, active or former
* History of ethambutol or synthetic antimalarial drug consumption
* History of chemotherapy
* Active and regular use of drugs
* non-weaned chronic alcoholism
* contra indication to MRI
* diabetes
* cognitive disorders (MoCA<26)
* non covered by health insurance
* patient under legal protection
* pregnant or breast-feeding woman
* Non inclusion criteria for control patients: known HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients infected for at least 10 years with undetectable viral load, selected among infectious disease outpatients (consecutive exhaustive recruitment)
  non HIV patients matched for age and gender
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
thickness of the RNFL and the RCGs measured by spectral domain OCT, between the two groups of patients | one day of examinations

CONTACTS AND LOCATIONS:
Overall Officials: Cédric LAMIREL, Dr, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild; Philippe GIRARD, Dr, Principal Investigator — Institut Mutualiste Montsouris; Antoine MOULIGNIE, Dr, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation OPH A de Rothschild, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Lamirel C, Valin N, Savatovsky J, Lescure FX, Alonso AS, Girard P, Vincensini JP, Girard PM, Salomon L, Cochereau I, Moulignier A. Absence of peripapillary retinal nerve-fiber-layer thinning in combined antiretroviral therapy-treated, well-sustained aviremic persons living with HIV. PLoS One. 2020 Mar 10;15(3):e0229977. doi: 10.1371/journal.pone.0229977. eCollection 2020. PMID 32155200